CLINICAL TRIAL: NCT03266887
Title: Association of Pre-diagnostic Vitamin D Levels and Survival in Older Individuals With Cancer
Brief Title: Vitamin D Levels and Survival in Cancer Patients
Status: Completed | Type: Observational
Sponsor: Icelandic Heart Association (Other)
Collaborators: University of Iceland (Other)
Responsible Party: Sponsor
Other Study IDs: HI14010102
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Using the population-based data sources in Iceland and the well-characterized AGES-Reykjavik cohort, our overarching aims are on exploring whether pre-diagnostic serum levels of 25-hydroxyvitamin D (25(OH)D) among older individuals living in Iceland were associated with survival after cancer diagnosis. We also wanted to assess the risk of being diagnosed with cancer in association with 25(OH)D levels. In this population living just south of the arctic circle, vitamin D levels largely depend on dietary- and supplemental sources.

ELIGIBILITY:
Inclusion Criteria:

To be part of the AGES-Reykjavik Study, initiated between 2002 and 2006.

Exclusion Criteria:

Diagnosed with cancer at study entry

Ages: 66 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: In 1967, all 30,795 men and women living in the capital area of Iceland and born between 1907 and 1935 were invited by the Icelandic Heart Association to join a prospective cohort study. Approximately 19,000 attended the clinic at least once and became participants of the Reykjavik Study. Subsequently, in 2002, a random sample of the cohort comprising 5,764 men and women who were still alive in Iceland and aged 66 to 96 years entered the Ages Gene/Environment Susceptibility (AGES) - Reykjavik Study (20). Serum 25(OH)D was measured in 5,519 of all 5,764 (96%) participants at study entry in year 2002 through 2006.
Sampling Method: Probability Sample
Enrollment: 5764 (Actual)
Dates: Start 2002-01-01 (Actual); Primary Completion 2006-12-30 (Actual); Study Completion 2006-12-30 (Actual)

PRIMARY OUTCOMES:
Overall mortality among cancer patients | Patients were followed from date of diagnosis since 2002 until death or censored at end of the follow-up (December 31, 2014)
  We tested the association between pre-diagnostic 25(OH)D levels and total survival

SECONDARY OUTCOMES:
Cancer-specific mortality among cancer patients | Patients were followed from date of diagnosis since 2002 until death or censored at end of the follow-up (December 31, 2014)
  We tested the association between pre-diagnostic 25(OH)D levels and cancer survival

OTHER OUTCOMES:
Pre-diagnostic 25(OH)D levels and cancer risk | Participants without cancer were followed from the study entry since 2002 until cancer diagnosis, death or end of the observation period whichever occurred first (December 31, 2014)
  We tested the association between pre-diagnostic 25(OH)D levels and risk of being diagnosed with cancer

REFERENCES:
- See also: Age, Gene/Environment Susceptibility-Reykjavik Study: Multidisciplinary Applied Phenomics — https://www.ncbi.nlm.nih.gov/pubmed?term=American+journal+of+epidemiology%5BJour%5D+AND+Harris+TB%5Bfirst+author%5D+AND+Age%2C+Gene/Environment+Susceptibility%E2%80%93Reykjavik+Study%3A+Multidisciplinary+Applied+Phenomics&TransSchema=title&cmd=detailssearch